CLINICAL TRIAL: NCT06782750
Title: The EFFECT of PHYSIOTHERAPY on CORPUS CALLOSUM VOLUME in STROKE PATIENTS
Brief Title: EFFECT of PHYSIOTHERAPY in STROKE
Status: Completed | Type: Observational
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Songül Bağlan Yentür, Head of Physiotherapy and Rehabilitatrion, Firat University
Other Study IDs: 250963
Record Dates: First submitted 2024-12-06; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-12

CONDITIONS: Stroke
Keywords: Corpus Callosum; Hemiplegia; Physiotherapy; Stroke
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hemiplegic patients: Patients had unilateral hemiplegia, practiced a rehabilitation program at the Physical Medicine and Rehabilitation Clinic of Firat University, and had no other neurological disease, were selected for the right and left groups.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Traditional physiotherapy treatment was applied 5 days in a week, 1 hour in a day for 6 weeks.

SUMMARY:
The study was aimed to determine the volumetric change in the corpus callosum after the rehabilitation program in patients with stroke. A total of 42 patients (22 males, 20 females), 21 right hemiplegic and 21 left hemiplegic patients with unilateral hemiplegia were enrolled in the rehabilitation program. Traditional physiotherapy treatment was applied 5 days in a week, 1 hour in a day for 6 weeks. The corpus callosum volumes were measured and evaluated on Magnetic Resonance Imaging (MRI) images before and after the treatment.

DETAILED DESCRIPTION:
Physical therapy after stroke contributes to the physical and social recovery of the paralyzed person. Corpus callosum is the commissural fibers consisting of white matter connecting the cortical areas between hemispheres. Its main function is to provide information exchange and coordination by establishing interhemispheric connections between areas in the right and left hemispheres. Inactivity and decreased physical activity may cause a decrease in the volume of the corpus callosum in patients with stroke. It was aimed to determine the volumetric change in the corpus callosum after the rehabilitation program in patients with stroke. A total of 42 patients (22 males, 20 females), 21 right hemiplegic and 21 left hemiplegic patients with unilateral hemiplegia were enrolled in the rehabilitation program. Traditional physiotherapy treatment was applied 5 days in a week, 1 hour in a day for 6 weeks. The corpus callosum volumes were measured and evaluated on Magnetic Resonance Imaging (MRI) images before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stroke
* Patients had unilateral hemiplegia
* Patients practiced a rehabilitation program at the Physical Medicine and Rehabilitation

Exclusion Criteria:

* Patients had other neurological disease
* Patients had mental disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with stroke, had unilateral hemiplegia, practiced a rehabilitation program at the Physical Medicine and Rehabilitation Clinic of XXX University, and had no other neurological disease, were selected for the right and left groups.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Corpus Callosum Volume | up to 2 weeks
  The measurements of the patients were evaluated on sagittal T2-weighted images. The slice thickness is 1.1 mm. Starting from the slice where the borders of the corpus callosum were clearly seen on the sagittal images, the circumference of the corpus callosum was marked on all sagittal slices where the borders of the corpus callosum were seen in consecutive slices.

CONTACTS AND LOCATIONS:
Overall Officials: Songul Baglan Yentur, Principal Investigator — Firat University
Locations (1):
- Firat University, Elâzığ, University, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No